CLINICAL TRIAL: NCT03597620
Title: An Investigator Initiated Open Label Study Evaluating the Efficacy and Tolerability of Application of Metaderm Product for the Treatment of Psoriasis
Brief Title: Evaluating the Efficacy and Tolerability of Application of Metaderm Product for the Treatment of Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Boni Elewski, Profesor and Chair, Department of Dermatology, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 180530
Record Dates: First submitted 2018-07-09; First posted 2018-07-24 (Actual); Results first posted 2022-10-03 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: 15 eligible patients will be enrolled. Patient will be treated for 12 weeks. There will be a total of five visits: screening, baseline, w4, w8 and w12. Metaderm cream will be applied topically twice a day to all active lesions. The metaderm scalp spray will be applied daily to the affected areas on the scalp. Patients will be provided with metaderm cleanser, can be use daily. For scalp psoriasis, patient will also use the shampoo Head & Shoulders formula with 1% Pyrithione Zinc as the active ingredient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nonsystemic Therapy + Herbal Anti-Inflammatory Treatment (HAT1) (Experimental): Patients who received HAT1 and were not on systemic treatment at time of enrollment. Metaderm cream will be applied topically twice a day to all active lesions. The metaderm scalp spray will be applied daily to the affected areas on the scalp.
  Interventions: Drug: Metaderm
- Systemic Therapy + Herbal Anti-Inflammatory Treatment (HAT1) (Experimental): Patients who received HAT1 and were on systemic treatment at time of enrollment. Metaderm cream will be applied topically twice a day to all active lesions. The metaderm scalp spray will be applied daily to the affected areas on the scalp.
  Interventions: Drug: Metaderm

INTERVENTIONS:
Drug: Metaderm — Metaderm cream and spray will be apply to subjects scalp and body.

SUMMARY:
Psoriasis vulgaris is a common inflammatory condition of the skin that results in well-demarcated, scaly, erythematous, itchy plaques. In the United States, psoriasis remains a common, immune-mediated disease, affecting 7.4 million adults. Often topical prescription medications are used as first line treatment for moderate psoriasis. Some topical medications have side effects and risk with long time use, thus not ideal for extensive and indefinite amount of time. Conversely, over- the-counter emollient treatments are readily available, safe and potentially efficacious. This study is design to test the safety and efficacy of topical application of the Metaderm product cream. The Metaderm cream is non-prescription, natural product.

ELIGIBILITY:
Inclusion Criteria for patients with plaque psoriasis 3-10% BSA

Subjects must satisfy the following criteria to be enrolled in the study:

1. Must be in general good health (except for disease under study) as judged by the Investigator, based on medical history, physical examination, clinical laboratories, and urinalysis. (NOTE: The definition of good health means a subject does not have uncontrolled significant co-morbid conditions).
2. Patients 18 and older
3. Give written informed consent prior to any study procedures being conducted, and candidates will authorize the release and use of protected health information (PHI)
4. Be willing and consent to having photos taken of their skin
5. Diagnosis of chronic plaque psoriasis that has been present for at least 6 months prior to baseline
6. Plaque psoriasis involving at least 3-10% of the patient's body surface area
7. Must have discontinued all systemic therapies for the treatment of psoriasis or psoriatic arthritis at least 4 weeks or 5 half-lives, and biologics 6 months) prior to baseline visit
8. Must have discontinued all topical therapies for the treatment of psoriasis at least 2 weeks prior to baseline visit
9. Subjects must have discontinued UV therapy at least 2 weeks prior to baseline and PUVA at least 4 weeks prior to baseline.
10. Subjects must be in good general health without significant uncontrolled comorbidities, other than psoriasis, as determined by the investigator based on exam findings, medical history, and clinical laboratories. Patients with stable mild renal insufficiency are eligible for enrolling in this trial.
11. Females of childbearing potential must use an approved birth control method while receiving treatment and for 28 days following the investigational product and there must be a documented negative pregnancy tests prior to initiating treatment. Approved birth control methods include hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring), intrauterine device, tubal ligation (tying your tubes), partners vasectomy, or male or female condoms that are not made of natural materials PLUS a diaphragm with spermicide, cervical cap with spermicide, or a contraceptive sponge with spermicide. Females not of child bearing potential are defined as being at least 1 year postmenopausal or surgically sterile (bilateral tubal ligation, bilateral oophorectomy and/or hysterectomy).

Inclusion Criteria with stable dose of biologic treatment and have plaque psoriasis 3-10 %BSA

Subjects must satisfy the following criteria to be enrolled in the study:

1. Must be in general good health (except for disease under study) as judged by the Investigator, based on medical history, physical examination, clinical laboratories, and urinalysis. (NOTE: The definition of good health means a subject does not have uncontrolled significant co-morbid conditions).
2. Patients 18 and older
3. Give written informed consent prior to any study procedures being conducted, and candidates will authorize the release and use of protected health information (PHI)
4. Be willing and consent to having photos taken of their skin
5. Diagnosis of chronic plaque psoriasis that has been present for at least 6 months prior to baseline
6. Stable dose of biologic therapy for the last 6 months prior to screening visit
7. Plaque psoriasis involving at least 3-10% of the patient's body surface area
8. Must have discontinued all topical therapies for the treatment of psoriasis at least 2 weeks prior to baseline visit
9. Subjects must have discontinued UV therapy at least 2 weeks prior to baseline and PUVA at least 4 weeks prior to baseline.
10. Subjects must be in good general health without significant uncontrolled comorbidities, other than psoriasis, as determined by the investigator based on exam findings, medical history, and clinical laboratories. Patients with stable mild renal insufficiency are eligible for enrolling in this trial.
11. Females of childbearing potential must use an approved birth control method while receiving treatment and for 28 days following the investigational product and there must be a documented negative pregnancy tests prior to initiating treatment. Approved birth control methods include hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring), intrauterine device, tubal ligation (tying your tubes), partners vasectomy, or male or female condoms that are not made of natural materials PLUS a diaphragm with spermicide, cervical cap with spermicide, or a contraceptive sponge with spermicide. Females not of child bearing potential are defined as being at least 1 year postmenopausal or surgically sterile (bilateral tubal ligation, bilateral oophorectomy and/or hysterectomy).

Inclusion Criteria for patients with scalp psoriasis

Subjects must satisfy the following criteria to be enrolled in the study:

1. Must be in general good health (except for disease under study) as judged by the Investigator, based on medical history, physical examination, clinical laboratories, and urinalysis. (NOTE: The definition of good health means a subject does not have uncontrolled significant co-morbid conditions).
2. Patients 18 and older
3. Give written informed consent prior to any study procedures being conducted, and candidates will authorize the release and use of protected health information (PHI)
4. Be willing and consent to having photos taken of their skin
5. Diagnosis of chronic plaque psoriasis that has been present for at least 6 months prior to baseline
6. Plaque psoriasis involving the scalp
7. Body plaque psoriasis cannot exceed 10 %BSA
8. Must have discontinued all systemic therapies for the treatment of psoriasis or psoriatic arthritis at least 4 weeks or 5 half-lives, and biologics 6 months) prior to baseline visit
9. Must have discontinued all topical therapies for the treatment of psoriasis at least 2 weeks prior to baseline visit
10. Subjects must have discontinued UV therapy at least 2 weeks prior to baseline and PUVA at least 4 weeks prior to baseline.
11. Subjects must be in good general health without significant uncontrolled comorbidities, other than psoriasis, as determined by the investigator based on exam findings, medical history, and clinical laboratories. Patients with stable mild renal insufficiency are eligible for enrolling in this trial.
12. Females of childbearing potential must use an approved birth control method while receiving treatment and for 28 days following the investigational product and there must be a documented negative pregnancy tests prior to initiating treatment. Approved birth control methods include hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring), intrauterine device, tubal ligation (tying your tubes), partners vasectomy, or male or female condoms that are not made of natural materials PLUS a diaphragm with spermicide, cervical cap with spermicide, or a contraceptive sponge with spermicide. Females not of child bearing potential are defined as being at least 1 year postmenopausal or surgically sterile (bilateral tubal ligation, bilateral oophorectomy and/or hysterectomy).

    Exclusion Criteria

    The presence of any of the following will exclude a subject from enrollment:
13. Other than disease under study, any clinically significant (as determined by the Investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is currently uncontrolled.
14. Any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study.
15. Prior history of suicide attempt at any time in the subject's life time prior to screening or randomization, or major psychiatric illness requiring hospitalization within the last 3 years.
16. Pregnant or breast feeding.
17. Active substance abuse or a history of substance abuse within 6 months prior to Screening.
18. Use of any investigational drug within 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamic half lives, if known (whichever is longer).
19. Prior treatment with the investigational product
20. Unable to comply with the protocol (as defined by the Investigator; i.e. drug or alcohol abuse or history of noncompliance)
21. Any other dermatologic conditions that prohibit or confound the ability of the investigator to interpret skin and/or nail exam findings.
22. Patients who will be unable to avoid the use of systemic steroids, excluding intranasal or inhaled steroids that will be permitted, for the duration of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2022-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boni Elewski, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Dermatology at the Whitaker Clinic, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nonsystemic Therapy + Herbal Anti-Inflammatory Treatment (HAT1): Participants who received HAT1 treatment and were not on systemic treatment at time of enrollment
- Systemic Therapy + Herbal Anti-Inflammatory Treatment: Participants who received HAT1 treatment and were on systemic treatment at time of enrollment.
Period: Overall Study
Arm/Group | Nonsystemic Therapy + Herbal Anti-Inflammatory Treatment (HAT1) | Systemic Therapy + Herbal Anti-Inflammatory Treatment
Started | 6 | 5
Completed | 4 | 5
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Systemic Therapy + Herbal Anti-Inflammatory Treatment (HAT1): Participants who received HAT1 treatment and were on systemic treatment at time of enrollment
- Total: Total of all reporting groups
Arm/Group | Nonsystemic Therapy + Herbal Anti-Inflammatory Treatment (HAT1) | Systemic Therapy + Herbal Anti-Inflammatory Treatment (HAT1) | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Efficacy as Measured by the Mean Percentage Change in the Product of Static Physician Global Assessment (sPGA) and Body Surface Area (BSA).
Description: The sPGA is the physician's global assessment of the subjects plaque psoriasis at a given time point. Plaques are assessed for induration, erythema, and scaling and an overall rating of plaque psoriasis severity is gen using the anchors of clear (0), minimal (1), mild (2), moderate (3), severe (4), or very severe (5).
  The BSA is the amount of body surface area affected by a disease. In this, the head represents 10% of the body, the upper extremities 20%, the trunk 30%, and the lower extremities 40%.
  These assessments will be combined by multiplying the numerical outcomes of the sPGA and BSA assessments to form a result. The mean change in this result will then be reported as the efficacy outcome. The data was all inclusive and not divided out by arm.
Time Frame: Baseline to Week 12
Measure: Mean (Standard Deviation); unit: percentage of change in sPGAxBSAscore
Groups:
- Nonsystemic Therapy+ Herbal Anti-Inflammatory Treatment (HAT1): Participants who received HAT1 and were not on systemic treatment at time of enrollment
- Systemic Therapy + Herbal Anti-Inflammatory Treatment (HAT1): Participants who received HAT1 and were on systemic treatment at time of enrollment
Arm/Group | Nonsystemic Therapy+ Herbal Anti-Inflammatory Treatment (HAT1) | Systemic Therapy + Herbal Anti-Inflammatory Treatment (HAT1)
Number analyzed (Participants) | 6 | 5
percentage of change in sPGAxBSAscore | 53.06 (40.01) | 65.6 (19.40)

2. Secondary Outcome: Efficacy as Measured by the Percentage Change in the DLQI. (Dermatology Quality of Life Index).
Description: The dermatology quality of life index (DLQI) is a simple, subject administered, 10 question validated, quality of life questionnaire that cover 6 domains including symptoms and feelings, daily activities, leisure, work, and school, personal relationships, and treatment. Response categories include "not at all", "a lot", and "very much", with corresponding score of 1, 2, and 3, respectively, and unanswered ("not relevant") responses scored as "0." The recall period is "over the last week," totals range from 0 to 30 (less to more impairment), and a 5-point change from baseline is considered clinically relevant. The data was all inclusive and not divided out by arm.
Time Frame: Baseline to Week 12
Measure: Mean (Standard Deviation); unit: percentage change for DLQI
Groups:
- Nonsystemic Therapy + Herbal Anti-Inflammatory Treatment (HAT1): Participants who received HAT1 and were not on systemic treatment at time of enrollment
Arm/Group | Nonsystemic Therapy + Herbal Anti-Inflammatory Treatment (HAT1) | Systemic Therapy + Herbal Anti-Inflammatory Treatment (HAT1)
Number analyzed (Participants) | 6 | 5
percentage change for DLQI | 52.88 (45.66) | 17.82 (36.68)

ADVERSE EVENTS:
Time Frame: Adverse event data was collect over the life of the trial (12 weeks).
Arm/Group | Nonsystemic Therapy + Herbal Anti-Inflammatory Treatment (HAT1) | Systemic Therapy + Herbal Anti-Inflammatory Treatment (HAT1)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5

LIMITATIONS AND CAVEATS:
This study is limited by the absence of a vehicle-controlled arm and its small number of patients. The addition of patients on systemic medications may also confound the results of the study. The results would benefit from a larger cohort and longer study duration to assess for long term efficacy and adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT03597620/Prot_SAP_000.pdf